CLINICAL TRIAL: NCT01073891
Title: Single-dose, Open-label, Randomized, Non-blinded, Three-fold Crossover Study in Healthy Subjects to Compare the Bioavailability of Moxifloxacin (BAY12-8039) 400 mg Tablet and 400 mg Oral Suspension Under Fasting Conditions, and to Investigate the Effect of Food on the Bioavailability of 400 mg Suspension.
Brief Title: Bioavailability, Food Effect and Safety, Tolerability of a New Oral Suspension in Comparison to the Marketed Moxifloxacin Tablet in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14413; 2009-017070-21 (EudraCT Number)
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Bioavailability; Food effect; Oral liquid formulation
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator)
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)
- Arm 2 (Experimental)
  Interventions: Drug: Moxifloxacin (BAY12-8039)
- Arm 3 (Experimental)
  Interventions: Drug: Moxifloxacin (BAY12-8039)

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — Single oral dose of moxifloxacin (Avelox, BAY12-8039) IR (immediate release) tablet 400 mg under fasting conditions
  Arms: Arm 1
Drug: Moxifloxacin (BAY12-8039) — Single oral dose of moxifloxacin (BAY12-8039) oral suspension 400 mg under fasting conditions
  Arms: Arm 2
Drug: Moxifloxacin (BAY12-8039) — Single oral dose of moxifloxacin (BAY12-8039) oral suspension 400 mg under fed conditions
  Arms: Arm 3

SUMMARY:
The purpose of this study is to describe the pharmacokinetics of a new oral liquid moxifloxacin formulation and the influence of concommitant food intake on the pharmacokinetics in healthy adults compared to the marketed oral tablet. Pharmacokinetics is to see how the body absorbs, distributes and gets rid of the study drug. The absorption of the drug administered in a different dosage form may be altered due to the influence of different excipients used. The safety of moxifloxacin when administered as an oral liquid formulation will also be looked at. Results from this study will be used to guide dosing strategies of the larger clinical trial planned for children.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects;
* Age: 18 to 55 years (inclusive)
* Body mass index (BMI): above/equal 18 and below/equal 30 kg/m²;
* Women of childbearing age must have a negative pregnancy test and must use adequate contraception throughout the study and for 4 weeks afterwards

Exclusion Criteria:

* Clinically relevant findings in the ECG
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Known hypersensitivity to moxifloxacin, other quinolones or to any of the excipients
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Relevant diseases within the last 4 weeks prior to the first study drug administration
* Febrile illness within 1 week before the first study drug administration
* Patients with a history of tendon disease/disorder related to quinolone treatment.
* Congenital or documented acquired QT prolongation
* Regular use of medicines (with the exception of contraceptives)
* Pregnancy or lactation
* Regular use of therapeutic or recreational drugs
* Smoking more than 25 cigarettes daily
* Regular daily consumption of more than 500 mL of usual beer or the equivalent quantity of approximately 20 g of alcohol in another form
* Suspicion of drug or alcohol abuse
* Special diets preventing the subjects from eating the standard meals during the study
* Regular daily consumption of more than 1 L of xanthin-containing beverages
* Donation of more than 100 mL of blood within 4 weeks before the first study drug administration or of approximately 500 mL in the preceding 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC) of Moxifloxacin after a Single Dose | 0 hour (pre-dose), 15, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours postdose
  AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC is defined as area under concentration versus time curve from time 0 (pre-dose) to extrapolated infinite time. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Maximum Observed Drug Concentration (Cmax) of Moxifloxacin after a Single Dose | 0 hour (pre-dose), 15, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours postdose
  Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to Infinity Divided by Dose(AUC/D) of Moxifloxacin after a Single Dose | 0 hour (pre-dose), 15, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours postdose
  Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Maximum Observed Drug Concentration Adjusted by Dose (Cmax/D) of Moxifloxacin after a Single Dose | 0 hour (pre-dose), 15, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours postdose
  Geometric mean and percentage geometric coefficient of variation (%CV) were reported.

SECONDARY OUTCOMES:
Area Under the Concentration Versus Time Curve From Zero to Infinity Divided by Dose per Kilogram Body Weight (AUC,norm) of Moxifloxacin after a Single Dose | 0 hour (pre-dose), 15, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours postdose
  AUC is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption. AUCnorm is defined as AUC divided by dose per kg body weight. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Area Under the Concentration Versus Time Curve From Zero to Last Quantifiable Concentration [AUC(0-tlast)] of Moxifloxacin after a Single Dose | 0 hour (pre-dose), 15, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours postdose
  AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC(0-tlast) is defined as AUC from time zero to the last data point above the lower limit of quantification. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Maximum Observed Plasma Concentration Divided by Dose per Kilogram Body Weight (Cmax,norm) of Moxifloxacin after a Single Dose | 0 hour (pre-dose), 15, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours postdose
  Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. Cmax,norm is defined as Cmax divided by dose per kg body weight. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Mean Residence Time (MRT) of Moxifloxacin after a Single Dose | 0 hour (pre-dose), 15, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours postdose
  MRT is an average duration of the drug in the body, and is expressed in hours. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Time to Reach Maximum Drug Concentration in Plasma (tmax) of Moxifloxacin after a Single Dose | 0 hour (pre-dose), 15, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours postdose
  tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Terminal Half Life Associated With the Terminal Slope (t1/2) of Moxifloxacin after a Single Dose | 0 hour (pre-dose), 15, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours postdose
  Half life associated with terminal slope refers to the elimination of the drug. It is the time taken for the blood plasma concentration to reach half the concentration in the terminal phase of elimination. It is expressed in hours and derived from the terminal slope of the concentration versus time curve. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.
Apparent Oral Clearance (CL/F) of Moxifloxacin after a Single Dose | 0 hour (pre-dose), 15, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours postdose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Geometric mean and percentage geometric coefficient of variation (%CV) were reported.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Wuppertal, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/